CLINICAL TRIAL: NCT05377840
Title: Effect Cognitive Behavioral Therapy (CBT) in the Treatment of Anxiety and Depression in Patients With Inflammatory Bowel Disease
Brief Title: Use of Psychologist-administered Cognitive Behavioral Therapy (CBT) or Self-administered CBT for the Treatment of Anxiety and/or Depression in Inflammatory Bowel Disease (IBD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Crohn's & Colitis Foundation of America (CCFA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000031323; 878888 (Other Grant/Funding Number: Crohn's & Colitis Foundation of America (CCFA))
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease; Ulcerative Colitis (UC)
Keywords: anxiety, depression
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: In this prospective, single center, randomized treatment study, participants will be screening for anxiety and depression in an inflammatory bowel disease population (Crohn's disease and ulcerative colitis) using the Generalized Anxiety Disorder (GAD) questionnaire and the Patient Health Questionnaire (PHQ). Subjects with GAD scores of ≥8 will be considered to have anxiety and those with a PHQ score of ≥10 will be considered to have depression. All subjects with screening questionnaire scores positive for anxiety or depression will be randomized to treatment with either psychologist-administered or self-administered cognitive behavioral therapy (CBT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychologist-administered Cognitive Behavioral Therapy (Active Comparator): Participants in this arm will participate in psychologist-administered CBT to assess the impact it will have on anxiety or depression among patients with inflammatory bowel disease
  Interventions: Behavioral: Psychologist-administered Cognitive Behavioral Therapy
- Self-administered Cognitive Behavioral Therapy (Experimental): Participants in this arm will be given a patient education book that teaches how to self-administer cognitive behavioral therapy to assess the impact it will have on anxiety or depression among patients with inflammatory bowel disease
  Interventions: Behavioral: Self-Administered Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Psychologist-administered Cognitive Behavioral Therapy — CBT is a combined psycho-social intervention that aims to improve overall mental health focusing on developing coping strategies. For psychologist-administered CBT: Participants will have individual weekly sessions (virtually) lasting 60 minutes each over an 8-week period with 1 follow-up maintenance session at week 12.
  Arms: Psychologist-administered Cognitive Behavioral Therapy
Behavioral: Self-Administered Cognitive Behavioral Therapy — CBT is a combined psycho-social intervention that aims to improve overall mental health focusing on developing coping strategies. For self-administered CBT: Participants will be given a book written for patients on CBT for IBD with instructions on how to self-administer CBT.
  Arms: Self-administered Cognitive Behavioral Therapy

SUMMARY:
This is a prospective, single center, randomized treatment study to assess if anxiety and depression in participants with IBD can be improved with CBT compared to those treated with SKY.

DETAILED DESCRIPTION:
This is a prospective, single center, randomized treatment study, where participants will be screened for anxiety and depression in an inflammatory bowel disease (Crohn's disease and ulcerative colitis) population using the Generalized Anxiety Disorder (GAD) questionnaire and the Patient Health Questionnaire (PHQ). Participants with GAD scores of ≥8 will be considered to have anxiety and those with a PHQ score of ≥10 will be considered to have depression. All participants with screening questionnaire scores positive for anxiety or depression will be randomized to treatment with either cognitive behavioral therapy (CBT) with a clinical psychologist (virtual visits) or CBT using a book written for IBD patients. The GAD and PHQ surveys will be repeated post treatment at weeks 6, 12 and 24. The primary objective of this study is to assess for an improvement in GAD and PHQ scores among subjects treated with CBT comparing 2 modalities of CBT. The secondary objectives are to assess for improvements in health-related quality of life, based on short IBD Questionnaire scores; assess for improvement in pain scores, based on the Brief Pain Inventory Short Form; and assess for improvement in fatigue scores based on the FACIT-Fatigue Scale, among subjects with poor scores at baseline following treatment with CBT.

ELIGIBILITY:
Inclusion Criteria:

* verified inflammatory bowel disease (Crohn's disease and ulcerative colitis)
* IBD patients on a stable treatment regimen with no evidence of active intestinal inflammation based on either normal c-reactive protein and/or fecal calprotectin, imaging studies, or endoscopy who meet the criteria for anxiety or depression based on the screening questionnaires
* subjects who have been on stable doses of anxiety and/or depression medications (defined as no dose adjustment in the prior 12 weeks) at the screening visit who meet the criteria for anxiety and/or depression based on screening questionnaires and are willing to stay on the same dose of these medications throughout the study duration
* may meet the criteria for both anxiety and depression and cohort assignment will be based on the survey with the highest scores suggesting more severe symptoms

Exclusion Criteria:

* declines to participate for the full duration of the study
* evidence of active intestinal inflammation based on an elevated c-reactive protein and/or fecal calprotectin, imaging studies or endoscopy
* non-English speaker
* any subject who expresses suicidal ideation or has severe mental illness as they will be taken to the emergency room for urgent psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in anxiety scores using the Generalized Anxiety Disorder-7 (GAD-7) questionnaire | baseline, week 6, week 12, week 24 and week 52
  Change from baseline in anxiety using GAD-7 compared to week 6, week 12 and week 24 (post treatment). Generalized Anxiety Disorder-7 questionnaire is a 7-item validated questionnaire used to screen for anxiety with a range of scores from 0-3. A cumulative score of ≥8 is considered positive for anxiety with lower scores indicating no or mild anxiety.
Change from baseline in depression scores using the Patient Health Questionnaire-9 (PHQ-9) | baseline, week 6, week 12, week 24, and week 52
  Change from baseline in depression using PHQ-9 compared to week 6, week 12 and week 24 (post treatment). PHQ-9 is a 9-item validated questionnaire used to screen for depression with a range of scores from 0-45. A cumulative score of ≥10 is considered positive with lower scores indicating no or mild anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Gaidos, MD, FACG, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391